CLINICAL TRIAL: NCT02641301
Title: Study of the Concentrations of Long Acting Morphine After Oral Absorption in Subjects Who Underwent Gastric Bypass (OBEMO 2)
Brief Title: Sustained-release Morphine Pharmacokinetics in Roux-en-Y Gastric Bypass Subjects
Acronym: OBEMO2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, MD, PhD, Hopital Lariboisière
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OBEMO2
Record Dates: First submitted 2015-12-14; First posted 2015-12-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Bypass Complications
Keywords: obesity; Roux-en-Y-gastric bypass; pharmacokinetics; Pain; morphine
MeSH Terms: conditions — Obesity; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects Roux-en-Y-gastric bypass (RYGB) (Experimental): Sustained release morphine sulfate, 30 mg
  Interventions: Drug: Sustained release morphine sulfate, 30 mg
- Control volunteers matched with RYGB (Active Comparator): Sustained release morphine sulfate, 30 mg
  Interventions: Drug: Sustained release morphine sulfate, 30 mg

INTERVENTIONS:
Drug: Sustained release morphine sulfate, 30 mg — A single oral administration of a capsule of sustained release morphine sulfate, 30 mg, on one day.
  Other Names: Code : 333 236-9 ; Access market authorisation 3400933323691

SUMMARY:
The purpose of this study is to determine whether sustained release morphine pharmacokinetics parameters in patients undergone roux-en-y gastric bypass (RYGB) differ from subjects who did not. Our hypothesis is that exposure is comparable. Indeed, in the Study OBEMO (Determinants of Oral Morphine Answer Among Obese Patients Before and After Gastric Bypass; NCT00943969) the investigators observed changes in pharmacokinetics parameters for immediate release morphine, probably due to an earlier absorption of the morphine, in agreement with the expected clinical effect of this formulation.

DETAILED DESCRIPTION:
This is an open label study with two arms: patients undergone roux-en-y gastric bypass and volunteers who did not matched by sex, age and Body Mass Index (BMI). In the pharmacokinetic visit the subject takes an oral administration of sustained release morphine, 30 mg, then 11 samples are collected during 12 hours.

ELIGIBILITY:
Inclusion Criteria:

RYGB Group (n=12) :

* Subjects who undergone RYGB for at least 24 months
* Stable weight since almost one year (or weight loss below 10kg over the last year)

Control group (n=12) :

* Volunteers subjects, matched for age, sex, and Body mass index
* No history of bariatric surgery

Same characteristics

* Subjects volunteers for the study
* Age 20-65 years
* Written consent

Exclusion Criteria:

* Known allergy to morphine or naloxone
* Patients not affiliated to the french social security system
* Subjects yet recruited in a study with remuneration
* Abnormalities in liver function Prothrombin ratio <70% and/ or aspartate transaminase > 5 times the usual values and/ or alanine aminotransferase >5 times the usual values and/ or in renal function (creatinine clearance Modification of Diet in Renal Disease (MDRD) < 60ml/ min
* Respiratory insufficiency defined by an oximetry below 90%
* Pregnancy and breastfeeding
* Use of drugs contra-indicated or not advised with morphine:
* Agonists-antagonists opioids ( buprenorphine, nalbuphine, pentazocine ), naltrexone
* Alcohol intake > 30g by day
* Cough medicine morphine-like ( dextromethorphan, noscapine, pholcodine )
* Codeine, ethylmorphine
* Other morphine agonist ( alfentanil, codeine, dextromoramide, dextropropoxyphene, dihydrocodeine, fentanyl, oxycodone, pethidin, phenoperidine, remifentanil, sufentanil, tramadol )
* Barbiturates, benzodiazepines
* Rifampicin

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Morphine area under the curve (AUC0-inf) after its oral administration according to the morphine concentration. | During the study visit: morphine concentration at time hour 0,5 ; hour 1; hour 1,5 ; hour 2; hour2,5; hour3; hour 4; hour 5; hour 6; hour 8; hour 12 after its oral administration

SECONDARY OUTCOMES:
Area under ther curve [AUC] of morphine-3-glucuronide, morphine-6-glucuronide | During the study visit: concentration at time hour 0,5 ; hour 1; hour 1,5 ; hour 2; hour2,5; hour3; hour 4; hour 5; hour 6; hour 8; hour 12 after morphine oral administration
Time of the maximum plasma concentration [Tmax] of morphine, morphine-3-glucuronide, morphine-6-glucuronide | During the study visit: concentrations at time hour 0,5 ; hour 1; hour 1,5 ; hour 2; hour2,5; hour3; hour 4; hour 5; hour 6; hour 8; hour 12 after morphine oral administration
Observed clearance [Cl/F] of morphine, morphine-3-glucuronide, morphine-6-glucuronide | During the study visit: concentrations at time 0,5h; 1h; 1,5h; 2h; 2,5h; 3h; 4h; 5h; 6h; 8h; 12h after morphine oral administration
  Blood samples gathered from hour 0,5 to hour 12 and urine sample gathered from the start to the end of the study visit.
Observed Volume of distribution [Vd / F] of morphine, morphine-3-glucuronide, morphine-6-glucuronide | During the study visit: concentrations at time hour 0,5 ; hour 1; hour 1,5 ; hour 2; hour2,5; hour3; hour 4; hour 5; hour 6; hour 8; hour 12 after morphine oral administration
Plasma Half-Life [T1 /2] of morphine, morphine-3-glucuronide, morphine-6-glucuronide | During the study visit: concentrations at time hour 0,5 ; hour 1; hour 1,5 ; hour 2; hour2,5; hour3; hour 4; hour 5; hour 6; hour 8; hour 12 after morphine oral administration
Maximum plasma concentration [Cmax] of morphine, morphine-3-glucuronide, morphine-6-glucuronide | During the study visit: concentrations at time hour 0,5 ; hour 1; hour 1,5 ; hour 2; hour2,5; hour3; hour 4; hour 5; hour 6; hour 8; hour 12 after morphine oral administration

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois JB Bergmann, MD, PhD, Study Director — Hopital Lariboisiere
Locations (2):
- France (2):
  - Therapeutic Research Unit, Department of Internal Medicine, Hospital Lariboisiere, Paris
  - Hopital Pitie Salpetriere, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finucane MM, Stevens GA, Cowan MJ, Danaei G, Lin JK, Paciorek CJ, Singh GM, Gutierrez HR, Lu Y, Bahalim AN, Farzadfar F, Riley LM, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Body Mass Index). National, regional, and global trends in body-mass index since 1980: systematic analysis of health examination surveys and epidemiological studies with 960 country-years and 9.1 million participants. Lancet. 2011 Feb 12;377(9765):557-67. doi: 10.1016/S0140-6736(10)62037-5. Epub 2011 Feb 3. PMID 21295846
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Padwal RS, Gabr RQ, Sharma AM, Langkaas LA, Birch DW, Karmali S, Brocks DR. Effect of gastric bypass surgery on the absorption and bioavailability of metformin. Diabetes Care. 2011 Jun;34(6):1295-300. doi: 10.2337/dc10-2140. Epub 2011 Apr 8. PMID 21478461
- [Background] Skottheim IB, Stormark K, Christensen H, Jakobsen GS, Hjelmesaeth J, Jenssen T, Reubsaet JL, Sandbu R, Asberg A. Significantly altered systemic exposure to atorvastatin acid following gastric bypass surgery in morbidly obese patients. Clin Pharmacol Ther. 2009 Sep;86(3):311-8. doi: 10.1038/clpt.2009.82. Epub 2009 Jun 3. PMID 19494810
- [Background] Hamad GG, Helsel JC, Perel JM, Kozak GM, McShea MC, Hughes C, Confer AL, Sit DK, McCloskey CA, Wisner KL. The effect of gastric bypass on the pharmacokinetics of serotonin reuptake inhibitors. Am J Psychiatry. 2012 Mar;169(3):256-63. doi: 10.1176/appi.ajp.2011.11050719. PMID 22407114
- [Background] Raebel MA, Newcomer SR, Reifler LM, Boudreau D, Elliott TE, DeBar L, Ahmed A, Pawloski PA, Fisher D, Donahoo WT, Bayliss EA. Chronic use of opioid medications before and after bariatric surgery. JAMA. 2013 Oct 2;310(13):1369-76. doi: 10.1001/jama.2013.278344. PMID 24084922
- [Background] Hasselstrom J, Sawe J. Morphine pharmacokinetics and metabolism in humans. Enterohepatic cycling and relative contribution of metabolites to active opioid concentrations. Clin Pharmacokinet. 1993 Apr;24(4):344-54. doi: 10.2165/00003088-199324040-00007. PMID 8491060
- [Background] Gourlay GK. Sustained relief of chronic pain. Pharmacokinetics of sustained release morphine. Clin Pharmacokinet. 1998 Sep;35(3):173-90. doi: 10.2165/00003088-199835030-00002. PMID 9784932
- [Background] Lloret-Linares C, Hirt D, Bardin C, Bouillot JL, Oppert JM, Poitou C, Chast F, Mouly S, Scherrmann JM, Bergmann JF, Decleves X. Effect of a Roux-en-Y gastric bypass on the pharmacokinetics of oral morphine using a population approach. Clin Pharmacokinet. 2014 Oct;53(10):919-30. doi: 10.1007/s40262-014-0163-0. PMID 25141973
- [Background] Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2011. Obes Surg. 2013 Apr;23(4):427-36. doi: 10.1007/s11695-012-0864-0. PMID 23338049
- [Background] Padwal R, Brocks D, Sharma AM. A systematic review of drug absorption following bariatric surgery and its theoretical implications. Obes Rev. 2010 Jan;11(1):41-50. doi: 10.1111/j.1467-789X.2009.00614.x. Epub 2009 Jun 2. PMID 19493300
- [Background] Skottheim IB, Jakobsen GS, Stormark K, Christensen H, Hjelmesaeth J, Jenssen T, Asberg A, Sandbu R. Significant increase in systemic exposure of atorvastatin after biliopancreatic diversion with duodenal switch. Clin Pharmacol Ther. 2010 Jun;87(6):699-705. doi: 10.1038/clpt.2010.32. Epub 2010 May 5. PMID 20445535
- [Background] Roberts DL, Dive C, Renehan AG. Biological mechanisms linking obesity and cancer risk: new perspectives. Annu Rev Med. 2010;61:301-16. doi: 10.1146/annurev.med.080708.082713. PMID 19824817
- [Background] Lotsch J, Weiss M, Ahne G, Kobal G, Geisslinger G. Pharmacokinetic modeling of M6G formation after oral administration of morphine in healthy volunteers. Anesthesiology. 1999 Apr;90(4):1026-38. doi: 10.1097/00000542-199904000-00016. PMID 10201674
- [Background] Kharasch ED, Hoffer C, Whittington D, Sheffels P. Role of P-glycoprotein in the intestinal absorption and clinical effects of morphine. Clin Pharmacol Ther. 2003 Dec;74(6):543-54. doi: 10.1016/j.clpt.2003.08.011. PMID 14663457